CLINICAL TRIAL: NCT01543711
Title: Long Term Follow-up of Persistent Pain, Sensory Disturbances and Lymphedema After Breast Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Kenneth Geving Andersen, MD, Rigshospitalet, Denmark
Other Study IDs: 2007-41-1530
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer; Pain; Post Operative Pain; Lymphedema; Neuropathy
Keywords: Breast cancer; persistent pain; neuropathic pain; lymphedema
MeSH Terms: conditions — Breast Neoplasms; Pain; Pain, Postoperative; Lymphedema; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer survivors: Women treated for breast cancer, without signs of recurrence or metastasis

SUMMARY:
Persistent pain, sensory disturbances, lymphedema and functional impairment are frequently occurring late effects of breast cancer treatment. The investigators have previously published data on 3253 women treated for breast cancer in Denmark in the period 2005-2006. Very few studies have examined how these late effects change in time. The aim of this study is to examine in a well defined patient population any change in the prevalence of persistent pain, sensory disturbances, lymphedema and functional impairment, as well as risk factor profile.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary breast cancer between 2005-2006
* Participated in a study in 2008

Exclusion Criteria:

* Recurrent or new primary cancer
* Metastatic cancer
* Reconstructive surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Woman treated for breast cancer in Denmark 2005-2006, and participated in the study in 2008
Sampling Method: Non-Probability Sample
Enrollment: 2411 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Prevalence of persistent pain | 6-7 years post operative
  Prevalence of pain in the breast area, axilla, side of chest or arm, as a yes/no variable
Prevalence of patients changing pain status from the 2008 survey | 6-7 years

SECONDARY OUTCOMES:
Prevalence of sensory disturbance | 6-7 years
Prevalence of self reported lymphedma | 6-7 years
Prevalence of functional impairment | 6-7 years
Risk factors associated for persistent pain, sensory disturbances, lymphedema or functional impairment | 6-7 years
Prevalence of patients changing status of sensory disturbances and self reported lymphedma | 6-7 years
Risk factors associated to changing status of sensory disturbances and lymphedema | 6-7 years post operative

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Geving Andersen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Derived] Mejdahl MK, Andersen KG, Gartner R, Kroman N, Kehlet H. Persistent pain and sensory disturbances after treatment for breast cancer: six year nationwide follow-up study. BMJ. 2013 Apr 11;346:f1865. doi: 10.1136/bmj.f1865. PMID 23580693